CLINICAL TRIAL: NCT01518036
Title: The Use of Norditropin® in Turner's Syndrome
Brief Title: Use of Somatropin in Turner Syndrome
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GHTUR/BPD/1
Record Dates: First submitted 2012-01-20; First posted 2012-01-25 (Estimated); Last update posted 2017-02-28 (Actual); Status verified 2017-02

CONDITIONS: Genetic Disorder; Turner Syndrome
MeSH Terms: conditions — Genetic Diseases, Inborn; Turner Syndrome | interventions — Human Growth Hormone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Low dose (Experimental)
  Interventions: Drug: somatropin
- High dose (Experimental)
  Interventions: Drug: somatropin

INTERVENTIONS:
Drug: somatropin — 2.9 IU/m^2/day. Administered as once daily subcutaneous injection until final height is reached
  Arms: Low dose
Drug: somatropin — 4.3 IU/m^2/day. Administered as once daily subcutaneous injection until final height is reached
  Arms: High dose

SUMMARY:
This trial is conducted in Europe. The aim of this trial is to study the dose-response relationship and effect of somatropin (Norditropin®) on final height in girls with Turner Syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Turner Syndrome
* Not previously treated with growth hormone or androgen
* Well-documented height over the previous 12 months
* Informed consent of parents (and child if appropriate)

Exclusion Criteria:

* Growth hormone (GH) deficiency based on a GH stimulation test

Ages: 2 Years to 11 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child
Enrollment: 57 (Actual)
Dates: Start 1987-09-14 (Actual); Primary Completion 2004-04-11 (Actual); Study Completion 2004-04-11 (Actual)

PRIMARY OUTCOMES:
Final height in cm

SECONDARY OUTCOMES:
Ratio between change in bone age and change in chronological age
Age at onset of puberty
Adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Crawley, United Kingdom

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com